CLINICAL TRIAL: NCT01525563
Title: Duphaston in Cycle Regularization: A Post-marketing, Prospective, Multicenter, Observational Study
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-282
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Irregular Menstrual Cycle
Keywords: Duphaston Study
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with irregular Menstrual cycle: Adult subjects with irregular menstrual cycle and can be treated with Duphaston as per locally approved label can be enrolled.

SUMMARY:
In India Duphaston is approved and widely used for the treatment of progesterone deficiencies such as for management of dysmenorrhea, endometriosis, secondary amenorrhea, irregular cycles, dysfunctional uterine bleeding, pre-menstrual syndrome, threatened and habitual abortion, infertility due to luteal insufficiency, as well as part of hormone replacement therapy. One Indian study reported normalization of the cycle in 91.6% of women with menstrual problems after three cycles of therapy with dydrogesterone 10 mg given from 11th to the 25th day of the menstrual cycle. The mean cycle duration during dydrogesterone therapy in this study was noted to be 28.8 days, in contrast to 17.9 days (in the polymenorrhea group) and 50.6 days (in the oligomenorrhea group) before therapy. Furthermore, dydrogesterone also decreased the amount and duration of menstrual bleeding in this study.

However, there are limited data regarding Duphaston's role in achieving cycle regularization from post-marketing settings. Moreover, it is not well-known if the effect of Duphaston therapy persists after cessation of treatment and whether the persistent effect, if any, is related to the duration of Duphaston therapy.

Hence, in this observational study, given that (based on previous clinical studies as mentioned above) Duphaston plays a role in menstrual irregularities treatment, the goal is to tease out the possible implications of such treatment in terms of treatment length and response pattern.

DETAILED DESCRIPTION:
Primary objective:

• To determine percentage of patients reporting a regular cycle (defined as cycle duration between 21 to 35 days, inclusive) at the end of treatment period.

Secondary objectives:

A. For all patients:

* To describe evolution of cycle duration from baseline to end of treatment by assessing mean cycle duration (in days) at baseline, separately in polymenorrhea, (i.e., cycle duration < 21 days) and oligomenorrhea (i.e., cycle duration > 35 days) groups, and at the end of treatment.
* To describe evolution of duration of menstrual bleeding from baseline to end of treatment by assessing mean duration of menstrual bleeding (in days) at baseline and at the end of treatment.
* To describe evolution of amount of menstrual bleeding from baseline to end of treatment, by assessing average number of pads changed per day at baseline and at the end of treatment.
* To describe evolution of pain during menstruation (on a 11 point Likert Scale where 0 means no pain and 10 means worst pain) ) from baseline to end of treatment, by assessing mean and standard deviation of pain scores at baseline and at the end of treatment.
* To describe overall patient satisfaction (on a 5 point Clinical Global Impression of Severity scale, where 1 = very dissatisfied, 2 = dissatisfied, 3 = somewhat satisfied, 4 = satisfied, 5 = very satisfied) at the end of treatment, by assessing percentages of patients in each category at the end of treatment.
* To describe overall clinical response (on a 7 point Clinical Global Impression of Severity scale, where 1 = Normal, not at all ill, 2 = Borderline mentally ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Most extremely ill) ) at the end of treatment by assessing percentages of patients in each category at the end of treatment.

B. For patients who had achieved regular cycle at the end of treatment:

* To determine the percentage of patients still experiencing regular cycle (i.e., duration 21-35 days, inclusive) at the end of follow up period, out of total number of patients who had achieved cycle regularization at the end of treatment period.
* To determine median time to relapse (defined as cycle duration < 21 days or > 35 days) during the follow up period, for patients who had achieved regular cycle at the end of treatment, using Kaplan Meier's method to graphically plot time after cessation of treatment versus percentage of patients still having regular cycles.
* To determine any correlation between treatment duration (number of cycles of Duphaston treatment received) and persistence of effect (number of months until when regular cycles are maintained after cessation of Duphaston therapy), using linear regression analysis model.
* To describe evolution of duration of menstrual bleeding from cessation of treatment to end follow up, by assessing mean duration of menstrual bleeding (in days) at end of treatment and at the end of follow up.
* To describe evolution of amount of menstrual bleeding from cessation of treatment to end follow up, by assessing average number of pads changed per day at end of treatment and at the end of follow up.
* To describe evolution of pain during menstruation (on a 11 point Likert Scale where 0 means no pain and 10 means worst pain) from cessation of treatment to end follow up, by assessing mean and standard deviation of pain scores at end of treatment and at the end of follow up.

ELIGIBILITY:
Inclusion Criteria

* Women aged 18 years or older
* Suffering from irregular menstrual cycle for at least 3 months and for whom the physician decides to prescribe Duphaston, in accordance with locally approved package insert
* Patients willing to sign written authorization to provide data for the study

Exclusion Criteria

* Patients having known hypersensitivity to the active ingredient or excipients
* Patients having known or suspected progesterone-dependent neoplasms
* Patients having vaginal bleeding of unknown etiology
* Patients taking oral contraceptives
* Pregnant and lactating patients
* Any other condition that precludes use of Duphaston in a particular patient, in accordance with the contraindication, precautions and special warnings listed in the locally approve package insert (for example, patients with history of liver disease, porphyria or depression)
* Patients not willing to sign written authorization for data release consent form

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with irregular menstrual cycle
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Hegde, MD-DCh, Study Director — Abbott
Locations (32):
- India (32):
  - Site Reference ID/Investigator# 69002, Ahmedabad
  - Site Reference ID/Investigator# 68995, Ahmedabad
  - Site Reference ID/Investigator# 68991, Ahmedabad
  - Site Reference ID/Investigator# 68990, Bangalore
  - Site Reference ID/Investigator# 69503, Banglore
  - Site Reference ID/Investigator# 69502, Banglore
  - Site Reference ID/Investigator# 69742, Bengaluru
  - Site Reference ID/Investigator# 69743, Bengaluru
  - Site Reference ID/Investigator# 69324, Chennai
  - Site Reference ID/Investigator# 68994, Chennai
  - Site Reference ID/Investigator# 68407, Chennai
  - Site Reference ID/Investigator# 68405, Delhi
  - Site Reference ID/Investigator# 68402, Delhi
  - Site Reference ID/Investigator# 69505, Hyderabad
  - Site Reference ID/Investigator# 69683, Hyderabad
  - Site Reference ID/Investigator# 69682, Hyderabad
  - Site Reference ID/Investigator# 69000, Hyderabad
  - Site Reference ID/Investigator# 69005, Jaipur
  - Site Reference ID/Investigator# 68410, Jaipur
  - Site Reference ID/Investigator# 68414, Jaipur
  - Site Reference ID/Investigator# 68999, Jaipur
  - Site Reference ID/Investigator# 73773, Mumbai
  - Site Reference ID/Investigator# 68993, Mumbai
  - Site Reference ID/Investigator# 69007, Mumbai
  - Site Reference ID/Investigator# 69004, Mumbai
  - Site Reference ID/Investigator# 69506, Mumbai
  - Site Reference ID/Investigator# 68996, Mumbai
  - Site Reference ID/Investigator# 69006, New Delhi
  - Site Reference ID/Investigator# 69009, Pune
  - Site Reference ID/Investigator# 69010, Pune
  - Site Reference ID/Investigator# 68412, Pune
  - Site Reference ID/Investigator# 68989, Pune

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With Irregular Menstrual Cycle
Started | 1000
End of Treatment | 910 (Only patients who had cycle regularization at end of treatment were allowed to continue.)
3 Months Follow-up | 838 (Only patients who had cycle regularization at end of treatment were allowed to continue.)
Completed | 788 (6 Months Follow-up)
Not Completed | 212

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 1000
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 29.2 (7.41)
Sex/Gender, Customized [Number; unit: participants] — All patients were female
  participants
    Female | 1000

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Reporting a Regular Cycle
Description: Regular cycle is defined as cycle duration between 21 to 35 days, inclusive at the end of treatment period.
Time Frame: 6 months
Population: Intent-to-Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Subjects With Irregular Menstrual Cycle: All patients who had received at least one dose of treatment and had at least one efficacy assessment to assess cycle regularization during the end of treatment period.
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
percentage of participants | 96.7 [95.5 to 97.9]

2. Secondary Outcome: Change in Cycle Duration (in Days) From Baseline to End of Treatment (EOT)
Description: The evolution of cycle duration from baseline to EOT was assessed by mean cycle duration (in days) at baseline, separately in polymenorrhea and oligomenorrhea groups, and at the EOT. The patients were included in polymenorrhea group in case the cycle duration at baseline was less than 21 days and in oligomenorrhea group in case the cycle duration at baseline was greater than 35 days.
Time Frame: 6 months
Population: All patients were assessed for overall reduction in cycle duration (910).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
Days
  Cycle duration at baseline | 44.73 (25.38)
  Cycle duration at EOT | 28.59 (7.61)
  change from baseline to EOT | -16.14 (24.04)

3. Secondary Outcome: Amount of Menstrual Bleeding From Baseline to End of Treatment
Description: Assessment of average number of pads changed per day at baseline and at the end of treatment (EOT).
Time Frame: 6 months
Population: The amount of menstrual bleeding (based on no. of pads used per day) was analyzed for all subjects completing EOT and change was noted from baseline to EOT
Measure: Mean (Standard Deviation); unit: pads/day
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
pads/day
  baseline amount of bleeding | 3.08 (1.26)
  EOT amount of bleeding | 2.63 (0.89)
  Change from baseline to EOT | -0.45 (1.20)

4. Secondary Outcome: Evolution of Pain During Menstruation From Baseline to End of Treatment
Description: The scores for pain during menstruation were recorded on 11-point Likert scale on baseline and end of treatment where 0 means no pain, and 10 means worst pain.
Time Frame: 6 months
Population: The scores for pain during menstruation were recorded on 11-point Likert scale on baseline for all enrolled subjects and end of treatment where 0 means no pain, and 10 means worst pain.
Measure: Number; unit: participants
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
participants
  No. of participants at Baseline (Scale 0-No Pain) | 139
  No. of participants EOT (Scale 0-No Pain) | 200
  No. of participants Baseline (Scale 10-Worst Pain) | 5
  No. of participants EOT (Scale 10-Worst Pain) | 0

5. Secondary Outcome: Overall Patient Satisfaction
Description: The overall patient satisfaction was recorded on a 5 point Clinical Global Impression of Severity scale, where 1 = very dissatisfied, 2 = dissatisfied, 3 = somewhat satisfied, 4 = satisfied, 5 = very satisfied).
Time Frame: 6 months
Population: Overall at the EOT, of 910 patients population the overall satisfaction was assessed
Measure: Number; unit: participants
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
participants
  EOT - Patient satisfaction (very satisfied - 5) | 282
  EOT - Patient satisfaction (satisfied - 4) | 532

6. Secondary Outcome: Evolution of Duration of Menstrual Bleeding From Baseline to End of Treatment
Description: To observe the evolution of duration of menstrual bleeding from baseline to end of treatment by assessing mean duration of menstrual bleeding (in days) at baseline and at the end of treatment.
Time Frame: 6 months
Population: To observe the evolution of duration of menstrual bleeding from baseline (all enrolled) to end of treatment by assessing mean duration of menstrual bleeding (in days) at baseline and at the end of treatment (EOT).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
Days
  duration of menstrual bleeding at baseline (days) | 4.99 (3.15)
  duration of menstrual bleeding at EOT (days) | 4.29 (1.38)

7. Secondary Outcome: Overall Clinical Response
Description: Overall response (on a 7 point Clinical Global Impression of Severity scale, where 1 = Normal, not at all ill, 2 = Borderline ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Most extremely ill) at the EOT by assessing percentages of patients in each category at the EOT.
Time Frame: 6 months
Population: Overall response (on a 7 point Clinical Global Impression of Severity scale, where 1 = Normal, not at all ill, 2 = Borderline ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Most extremely ill) at the EOT by assessing percentages of patients in each category at the EOT.
Measure: Number; unit: participants
Arm/Group | Subjects With Irregular Menstrual Cycle
Number analyzed (Participants) | 910
participants
  Overall Clinical Response EOT (Normal, not ill) | 851
  Overall Clinical Response EOT(Most extremely ill) | 0

ADVERSE EVENTS:
Time Frame: 6 months treatment duration + 6 months follow up period (15 months)
Description: The safety analysis set included all enrolled patients who satisfied all inclusion and exclusion criteria
Arm/Group | Subjects With Irregular Menstrual Cycle
Serious Adverse Events (participants affected / at risk) | 1/1000
Other Adverse Events (participants affected / at risk) | 3/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Irregular Menstrual Cycle (N=1000)
Appendicitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Irregular Menstrual Cycle (N=1000)
Hypersensitivity (Immune system disorders) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 1 (1)
Menstruation Irregular (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other